CLINICAL TRIAL: NCT01428544
Title: Special Drug Use Investigation (Retrospective) for Arixtra® (Fondaparinux) Venous Thromboembolism Treatment (Over 100kg)
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: 115490
Record Dates: First submitted 2011-09-01; First posted 2011-09-05 (Estimated); Last update posted 2015-07-15 (Estimated); Status verified 2015-07

CONDITIONS: Ataxia
MeSH Terms: conditions — Ataxia | interventions — Fondaparinux

STUDY DESIGN:
Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with VTE treated with fondaparinux: Patients with VTE treated with fondaparinux
  Interventions: Drug: Fondaparinux sodium

INTERVENTIONS:
Drug: Fondaparinux sodium — For patients whose body weight is 100 kg or more, fondaparinux is injected 10 mg subcutaneously once daily for treatment of acute pulmonary thromboembolism or acute deep venous thrombosis.

SUMMARY:
The purpose of this post-marketing surveillance study is to collect and assess information retrospectively on safety and effectiveness of fondaparinux injection in patients with venous thromboembolism (VTE) whose body weight is 100 kilograms (kg) or more, or to whom fondaparinux was injected 10 mg/day.

("Arixtra" is a trademark of the GlaxoSmithKline group of companies.)

ELIGIBILITY:
Inclusion Criteria:

* Patients with acute pulmonary thromboembolism or acute deep venous thrombosis
* Fondaparinux injection must be prescribed for the first time

Exclusion Criteria:

* Not applicable

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Japanese patients with acute pulmonary thromboembolism or acute deep venous thrombosis whose body weight is 100 kg or more, or to whom fondaparinux was injected 10 mg/day.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2012-03; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Number of patients with adverse drug reaction | 3 months
Number of patients with any serious adverse event | 3 months
Number of patients with any hemorrhagic adverse event | 3 months
Presence or absence of reoccurrence of VTE | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline